CLINICAL TRIAL: NCT04515537
Title: The Effect of Cyanophyta Aphanizomenon Flos-aquae (Stemregen), and Adipose Stroma Vascular Fraction (SVF) Either Individual or in Combination in Patient With Heart Failure
Brief Title: Cyanophyta Aphanizomenon Flos-aquae, and Adipose Stroma Vascular Fraction, in Heart Failure Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Española de Medicina Regenerativa y Terapia Celular (Other)
Collaborators: Clinica Castello 68 (Other)
Responsible Party: Sponsor
Other Study IDs: 13245
Record Dates: First submitted 2020-01-03; First posted 2020-08-17 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Congestive Heart Failure Chronic
Keywords: Heart Failure; Stem Cell; Stroma vascular fraction; AFA
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- conventional therapy plus AFA: Patient using conventional therapy plus Extract of the Cyanophyta Aphanizomenon Flos-aquae (AFA), for a period of 6 months
  Interventions: Dietary Supplement: Water-soluble Extract of the Cyanophyta Aphanizomenon Flos-aquae (AFA),
- conventional therapy plus SVF: Patient using conventional therapy plus aplication of stroma vascular fraction (SVF) from the adipose tissue, evaluted for period of 6 months
  Interventions: Procedure: Infiltrtion of SVf
- conventional therapy plus SVF and AFA: Patient using conventional therapy plus aplication of stroma vascular fraction (SVF) from the adipose tissue plus Extract of the Cyanophyta Aphanizomenon Flos-aquae (AFA), for a period of 6 months
  Interventions: Dietary Supplement: Water-soluble Extract of the Cyanophyta Aphanizomenon Flos-aquae (AFA),; Procedure: Infiltrtion of SVf

INTERVENTIONS:
Dietary Supplement: Water-soluble Extract of the Cyanophyta Aphanizomenon Flos-aquae (AFA), — Patient use 2 capsules 3 time a day by oral.
  Groups: conventional therapy plus AFA; conventional therapy plus SVF and AFA
Procedure: Infiltrtion of SVf — After filling up the informed consent Mini liposuction is performed under local anesthesia with klein solution, about 70 cc of dry fat tissue is suctioned and collagenase digestion is done with final centrifugation to obtain the SVF
  Groups: conventional therapy plus SVF; conventional therapy plus SVF and AFA

SUMMARY:
This study is a prospective, randomized, controlled trial to assess the efficacy of transplantation of autologous stroma vauscultar fraction and/or AFA in 15 patients with ischemic heart failure

DETAILED DESCRIPTION:
Stem cells therapy may be a choice therapy for advanced heart failure patients refractory to medical therapy, and a previous history of coronary artery diseases. In this study the investigators have evaluated consecutive 15 selected patients, the amelioration in failing heart NYHA class, hospitalization rate, echocardiographic left ventricle functionality, serum of Natriuretic peptide level and associated to reduction of angina after a treatment with stroma vascular fraction infusion y/or Stemregen capsule per oral.

ELIGIBILITY:
Inclusion Criteria:

* EF < 45 %
* NYHA 2 - 3

Exclusion Criteria:

* Acute coronary syndrome within last 6 weeks.
* Pregnancy
* FEV1 <20 %
* Cancer
* Any severe disease which could interfere with the treatment or the outcome
* Patient with immunodeficiency
* Candidate who are judged to be not applicable to this study by doctors.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 patients age from 35 to 80 yers old
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change NYHA functional class assessed with SAQ-7 -questionnaire | 6 month
  The improvement in patient's quality of life after 6 months of trial admission. The quality of life will be determined with Seattle Angina Questionnaire 7 (SAQ-7). Each domain has a score calculated on a scale of 0 (= worst health quality) to 100 (= best health quality)
Change of echocardiographic Parameters [ Time Frame: 0 and 6 months ] | 6 months
  Left Ventricular end-systolic volume index (LVESVI) Left Ventricular end-systolic dimension Left Ventricular end-diastolic volume Left Ventricular end-diastolic dimension. [ Time Frame: 6 months from trial admission]

SECONDARY OUTCOMES:
Change NYHA functional class assessed with SAQ-7 -questionnaire | 12 months
  The improvement in patient's quality of life after 12 months of trial admission. The quality of life will be determined with Seattle Angina Questionnaire 7 (SAQ-7). Each domain has a score calculated on a scale of 0 (= worst health quality) to 100 (= best health quality).
Change of echocardiographic Parameters [ Time Frame: 0 and 12 months ] | 12 months
  Left Ventricular end-systolic volume index (LVESVI) Left Ventricular end-systolic dimension Left Ventricular end-diastolic volume Left Ventricular end-diastolic dimension, [ Time Frame: 12 months from trial admission]

CONTACTS AND LOCATIONS:
Overall Officials: Miguel G Garber, MD, Principal Investigator — Healthy Longevity Clinic; Christian Drapeau, PhD, Study Director — Kalyagen
Locations (1):
- Clinca Castello 68, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 15 months to 3 years
Access Criteria: Undecided

REFERENCES:
- [Background] Sheu JJ, Lee MS, Wallace CG, Chen KH, Sung PH, Chua S, Lee FY, Chung SY, Chen YL, Li YC, Yip HK. Therapeutic effects of adipose derived fresh stromal vascular fraction-containing stem cells versus cultured adipose derived mesenchymal stem cells on rescuing heart function in rat after acute myocardial infarction. Am J Transl Res. 2019 Jan 15;11(1):67-86. eCollection 2019. PMID 30787970
- [Background] Premaratne GU, Ma LP, Fujita M, Lin X, Bollano E, Fu M. Stromal vascular fraction transplantation as an alternative therapy for ischemic heart failure: anti-inflammatory role. J Cardiothorac Surg. 2011 Mar 31;6:43. doi: 10.1186/1749-8090-6-43. PMID 21453457
- [Background] Kelm NQ, Beare JE, Yuan F, George M, Shofner CM, Keller BB, Hoying JB, LeBlanc AJ. Adipose-derived cells improve left ventricular diastolic function and increase microvascular perfusion in advanced age. PLoS One. 2018 Aug 24;13(8):e0202934. doi: 10.1371/journal.pone.0202934. eCollection 2018. PMID 30142193
- [Background] Leblanc AJ, Nguyen QT, Touroo JS, Aird AL, Chang RC, Ng CK, Hoying JB, Williams SK. Adipose-derived cell construct stabilizes heart function and increases microvascular perfusion in an established infarct. Stem Cells Transl Med. 2013 Nov;2(11):896-905. doi: 10.5966/sctm.2013-0046. Epub 2013 Oct 8. PMID 24106337
- [Background] Jensen GS, Hart AN, Zaske LA, Drapeau C, Gupta N, Schaeffer DJ, Cruickshank JA. Mobilization of human CD34+ CD133+ and CD34+ CD133(-) stem cells in vivo by consumption of an extract from Aphanizomenon flos-aquae--related to modulation of CXCR4 expression by an L-selectin ligand? Cardiovasc Revasc Med. 2007 Jul-Sep;8(3):189-202. doi: 10.1016/j.carrev.2007.03.004. PMID 17765649
- [Background] Hart AN, Zaske LA, Patterson KM, Drapeau C, Jensen GS. Natural killer cell activation and modulation of chemokine receptor profile in vitro by an extract from the cyanophyta Aphanizomenon flos-aquae. J Med Food. 2007 Sep;10(3):435-41. doi: 10.1089/jmf.2007.401. PMID 17887936